CLINICAL TRIAL: NCT02209389
Title: OctavaPink® For Dense Breast After Negative Mammography
Brief Title: OctavaPink for Women With Dense Breast After Negative Mammography
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Eventus Diagnostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: OctavaPink for Dense Breast
Record Dates: First submitted 2014-07-29; First posted 2014-08-05 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; cancer associated auto antibodies; breast cancer blood test
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Human plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Positive OctavaPink: Following a positive OctavaPink result, an MRI is performed and any additional testing (required by the MRI).
  Interventions: Device: MRI
- Negative OctavaPink - control: For any sample that is identified with a positive OctavaPink result, a negative sample from the same center, as close in time as possible, and of the same age decade, will be identified and recalled for an MRI and any additional testing (required by the MRI).
  MRI won't be performed to all negative OctavaPink results. Only one negative control will be assigned to each OctavaPink positive result.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — For any sample that is identified with a positive OctavaPink result, a negative sample from the same center, as close in time as possible, and of the same age decade, will be identified and will be recalled for an MRI and any additional testing if requested by doctor's (according to MRI's results).
  Other Names: Magnetic Resonance Imaging

SUMMARY:
The OctavaPink test is indicated as an adjunct to mammography for breast cancer screening in asymptomatic women for whom screening or diagnostic mammography findings are normal or benign (BIRADS assessment category 1 or 2) and breast tissue is dense (BIRADS composition/density 3 or 4). The device is intended to increase breast cancer detection in the described patient population. Based upon the result of OctavaPink, the patient will be further evaluated by their physician.

DETAILED DESCRIPTION:
This is a multicenter, prospective study containing 3 parts:

Part 1 consists of Part 1A (optimization/training) and Part 1B (evaluation/testing) as follows:

Part 1A will optimize the OctavaPink test for women with dense breast tissue, and will not affect the treatment of the participants. Part 1A is an internal part done by EventusDx and no statistical evaluation is needed.

Objectives: To optimize the OctavaPink test, with the target of ≥95% specificity and ≥70% sensitivity.

Part 1B will assess the properties of the OctavaPink test using cases and controls obtained via the same criteria as in Part 1A. The sensitivity and specificity of the OctavaPink test must be confirmed as sufficiently high in samples in which EventusDx is blind to case/control status before using the test to affect clinical management of patients.

Objectives:

(i) To obtain a sensitivity estimate ≥60% with 95% CI lower limit ≥50% in the whole group of cancer cases (DCIS, IDC and ILC); also to obtain a sensitivity estimate with the same properties in the subset of cases with invasive cancer (IDC and ILC).

(ii) To obtain a specificity estimate ≥90% in controls with 95% CI lower limit ≥85%.

Part 2 will examine the yield of cancer detection by MRI/biopsy among women who have a positive OctavaPink test result in the dense breast negative mammography population.

Objectives:

(i) To compare the yield of cancer detection via MRI/biopsy among women with a positive OctavaPink test versus a negative OctavaPink test result.

(ii) To estimate the proportion of patients who are positive for the test in the target population

Part 3 will assess sensitivity of OctavaPink test in an enriched population of women with dense breasts and negative mammography.

Objectives: To obtain an estimate of sensitivity in women with dense breast tissue and negative mammography that is broadly consistent with that found in the dense breast population (but not necessarily negative mammogram) in Parts 1A and 1B.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with dense breast tissue according to ACR criteria, (BIRADS composition/density 3 or 4), or with specific area of high density behind the nipple.
* Subject with current mammography BIRADS assessment category other than 3.
* Signed inform consent form.

Additional inclusion criteria for Part 1A and Part 1B cases and Part 3 cases

• Subjects with current biopsy/surgery proven breast cancer.

Additional inclusion criteria for Part 1A controls, Part 1B controls • Subjects with current negative mammography (BIRADS assessment category 1 or 2).

Additional inclusion criteria for Part 2

• Subjects with current negative mammography (BIRADS assessment category 1 or 2). All will perform an additional 1 year (12-18 months) up mammography to verify negative results.

Additional inclusion criteria for Part 3 • Enriched patient population - Subjects with current/recent (less than 12 months) negative mammography (BIRADS assessment category 1 or 2). Mammography evaluation can be performed after recruiting.

Exclusion Criteria:

* Previous or concurrent malignancies of any type except for basal cell carcinoma of the skin, squamous-cell carcinoma of the skin or cervical carcinoma in situ.
* Previous or current ADH, ALH, LCIS.
* Autoimmune disorders diagnosed subjects.
* Hematological malignancies.
* Subjects under active chemotherapy treatment or chemotherapy in the past 6 months.
* Steroid treatment in the past 3 months.
* Subject undergoing immunosuppressive treatments.
* Subject with current mammography BIRADS assessment category of 3.
* Pregnancy at time of recruitment.
* Doctor medical judgment that prohibits participation in the study.
* Participating in a parallel clinical study that involves drug treatment, or may influence the course of this clinical trial.

Additional exclusion criteria for Part 3

• Subjects with current mammography BIRADS assessment other than 1 or 2.

Ages: 30 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population for all parts of the protocol includes women above 30, who have had a mammography in the past 5-18 months, for which the result was negative (BIRADS assessment category 1 or 2), and on which they were defined as having dense breast tissue (BIRADS composition/density 3 or 4).
Sampling Method: Probability Sample
Enrollment: 1750 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Positive MRI as an approval for a positive OctavaPink test | Approximately two month following a positive Octava test

CONTACTS AND LOCATIONS:
Overall Officials: Edith Perez, Prof., Principal Investigator — Mayo Clinic, Jacksonville Florida USA
Locations (7):
- United States (2):
  - Detroit Clinical Research Center, Detroit, Michigan
  - MD Anderson cancer center, Houston, Texas
- Israel (4):
  - Shaarey Tzedek, Jerusalem
  - Shiba, Ramat Gan
  - Kaplan medical center, Rehovot
  - Sourasky medical center, Tel Aviv
- Fondazione Carlo ferri, Rome, Italy

REFERENCES:
- [Background] Yahalom G, Weiss D, Novikov I, Bevers TB, Radvanyi LG, Liu M, Piura B, Iacobelli S, Sandri MT, Cassano E, Allweis TM, Bitterman A, Engelman P, Vence LM, Rosenberg MM. An Antibody-based Blood Test Utilizing a Panel of Biomarkers as a New Method for Improved Breast Cancer Diagnosis. Biomark Cancer. 2013 Nov 19;5:71-80. doi: 10.4137/BIC.S13236. eCollection 2013. PMID 24324350